CLINICAL TRIAL: NCT00705835
Title: Vaccine Therapy of Prostate Cancer Patients With Recombinant Soluble Prostate-Specific Membrane Antigen (Rs-PSMA) Plus the Immunological Adjuvant Alhydrogel: A Trial Studying RsPMSA Doses
Brief Title: Vaccine Therapy of Prostate Cancer Patients With Recombinant Soluble Prostate-Specific Membrane Antigen (Rs-PSMA) Plus the Immunological Adjuvant Alhydrogel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: PSMA Development Corp, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-072
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Prostate Cancer
Keywords: Prostate; ALHYDROGEL; RS-PSMA
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (2):
- 1 (Experimental): This is an ascending, multiple dose study in up to 18 patients. As many as eight patients are planned at each of two dose levels, intrapatient dose escalation is not allowed. Six patients will start on 50μg rsPSMA +0.5 mg Alhydrogel® Weeks 1,2,3 and 7.
  Interventions: Biological: rsPSMA protein plus Alhydrogel® vaccine
- 2 (Experimental): This is an ascending, multiple dose study in up to 18 patients. As many as eight patients are planned at each of two dose levels, intrapatient dose escalation is not allowed. Eight patients will start on 250μg rsPSMA + 1.0 mg Alhydrogel Weeks 1,2,3 and 7
  Interventions: Biological: rsPSMA protein plus Alhydrogel® vaccine

INTERVENTIONS:
Biological: rsPSMA protein plus Alhydrogel® vaccine — The assigned dose of rsPSMA protein plus Alhydrogel® vaccine will be administered subcutaneously to random sites on the upper arm and upper leg at weekly intervals for 3 weeks. This will be followed by a 4-week break and then a fourth vaccination during week 7. The vaccination site will rotate to a different quadrant with each administration.

SUMMARY:
The purpose of this research is to help us study a vaccine treatment for patients with prostate cancer. A vaccine is a medicine that teaches the body to destroy harmful infections and other diseases, such as cancer. Your immune system is made up of many different types of cells which fight infection and disease in your body. A vaccine may stimulate the immune system to destroy the cancer cells. It may also help to slow the growth of the cancer. The vaccine is a solution given as an injection into or under the skin. It is made up of several parts. The first part is PSMA, a protein present in many cancers, especially prostate cancer. It is referred to as rsPSMA when made in a laboratory for this study and is mixed with a material called Alhydrogel® (aluminum hydroxide suspension) which helps the immune system to make more cancer-fighting cells.

ELIGIBILITY:
Inclusion Criteria:

* Non-castrate metastatic patients must have biochemically progressive disease as defined by serial changes in PSA (with a serum testosterone > or = to 180 ng/mL)following definitive primary therapy such as prostatectomy or radiation. Castrate metastatic patients must have biochemically progressive disease in the absence of radiographic evidence of disease progression with rising PSA values despite castrate (<50 ng/mL) levels of testosterone following an adequate course of hormonal therapy. An adequate course of hormonal therapy is treatment with an LH-RH analog (with or without an anti-androgen) or orchiectomy.
* Prostate cancer must be histologically confirmed by the Department of Pathology at MSKCC.
* Karnofsky performance status >70%.
* Patients must have adequate organ function as defined by:
* WBC > or = to 3000/mm3, neutrophils > or = to1000/mm3, platelet count > or = to l00,000 mm3
* Bilirubin <2.0 mg/dl
* Alkaline Phosphatase and SGOT <3.0 times the upper limit of normal
* Creatinine < or = to 2.0 mg/dl
* Hemoglobin >9.0 g/dl
* ALT <2.5 times the upper limit of normal
* Patients must be at least 18 years of age
* Expected survival must be >6 months
* Patients must sign informed consent.
* Non-castrate metastatic patients must have a serum testosterone >180 ng/mL.

Exclusion Criteria:

* Radiographic evidence of disease progression.
* Clinically significant cardiac disease (New York Heart Association Class III/IV or severe debilitating pulmonary disease).
* Active CNS or epidural tumor.
* An infection requiring antibiotic treatment.
* Lymphopenia defined by lymphocytes <1000/mm3.
* Cancer related pain requiring the use of opioid containing analgesics.
* Positive stool guaiac, excluding hemorrhoids or documented radiation-induced proctitis.
* Concurrent treatment with nutritional or herbal supplements (e.g., PC SPES or similar agents) which could potentially confound the interpretation of study results.
* History of an active secondary malignancy except for non-melanoma skin cancer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2003-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Is to investigate the safety and tolerability of treatment with increasing dose levels of rsPSMA protein when administered with the adjuvant Alhydrogel®. | conclusion of study

SECONDARY OUTCOMES:
To evaluate the immune response to increasing dose levels of rsPSMA protein. | conclusion of study
To study the pattern of change in PSA after vaccination. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Susan Slovin, MD,PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org